CLINICAL TRIAL: NCT04412343
Title: The Seniors COvid-19 Pandemic and Exercise Study: A Randomized Controlled Trial
Brief Title: The Seniors COvid-19 Pandemic and Exercise Study
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Victoria (Other)
Responsible Party: Principal Investigator, Mark Beauchamp, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H20-01515
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Well-Being (Psychological Flourishing); Depression; Quality of Life; Loneliness; Physical Activity; Social Identification; Physical Health
MeSH Terms: conditions — Depression; Motor Activity; Social Identification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: No experimenter or investigator expectancy effects as all assessment occurs online (i.e., online questionnaire). Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual group exercise (Experimental): Individuals in the (virtual) group-based exercise program, will have the opportunity to take part in (virtual) group exercise classes, delivered via videoconferencing, by experienced older adult exercise instructors. Personnel who analyze the data collected from the study are not aware of the treatment applied to any given group. Classes will be offered multiple days a week at 9am PST (12 noon EST), and will last approximately 50 minutes. Classes include a warm-up component, moderate intensity exercises as the core component of the class, and a cool-down. At the end of classes participants will have the opportunity to connect in small groups (videoconferencing breakout groups) to socially connect over a beverage (coffee, water) from their own homes. Participants in the group condition will also be sent, by mail, a program t-shirt to foster a sense of distinctiveness.
  Interventions: Behavioral: Virtual Group Intervention
- Personal exercise (Experimental): Each of the older adult instructors described above will also contribute to delivering pre-recorded exercise classes (involving the same exercises, intensity, music, and so forth as those described above for the group condition). However, in this instance, instructors will deliver those classes to each participant by referring to themselves as each participant's personal trainer/coach, with language directed to the individual and not the group. That is, no sense of 'groupness' or 'shared social identities/connectivity' will be primed. Also, participants in this condition will not have the opportunity to interact with other older adults after classes have ended and will not receive the same program t-shirts designed to foster a sense of group distinctiveness.
  Interventions: Behavioral: Personal Exercise Intervention
- Wait-list control (No Intervention): Those randomized to the wait-list control condition will go about their daily lives for the duration of the 12-week trial. They will be asked to complete the same questionnaires (and will be remunerated in the same way as those in the other two conditions via $10 per questionnaire completion). At the end of the 12-week trial, participants in this condition will have access to the personal exercise programming.

INTERVENTIONS:
Behavioral: Virtual Group Intervention — Participants will receive weekly exercise courses delivered virtually to a group of older adults. This intervention will last for 12 weeks. Participants in addition to participating in exercise will have designated time after each exercise class to socially connect. Participants in this condition will also receive a t-shirt.
  Arms: Virtual group exercise
Behavioral: Personal Exercise Intervention — Participants will receive weekly exercise courses delivered virtually. These classes will be pre-recorded so the individual can complete sessions at any time that is convenient for them.
  Arms: Personal exercise

SUMMARY:
The purpose of this study is to evaluate different types of exercise programs (virtual group-based exercise program; personal exercise program; wait-list control) across 12-weeks on the physical and mental health of older adults during the current Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years old
* be able to speak and read English
* one participant in the study per household (Spouses, significant others, or family members can take part in the exercise programs with the study participant; however, they will not be able to provide data and won't be remunerated for participating)
* not experience any contraindication which might prevent that person from participating in moderate-intensity physical activity.
* participants must be able to access the internet at home via a personal smartphone, tablet (e.g., ipad), or computer (device used must have camera capabilities)
* low active individuals (i.e., less than 150 minutes of moderate-to-vigorous physical activity per week)
* currently living in Canada

Exclusion Criteria:

* age of less than 65 years
* unable to read and speak in English
* inability to participate in moderate-to-vigorous physical activity (including a lack of ability to receive doctor's clearance for participating in physical activity)
* lack of internet access which does not allow them to access online materials
* device used to access the internet does not have a camera/video capabilities
* active individuals (e.g., participate in greater than 150 minutes of moderate-to-vigorous physical activity each week)
* living outside Canada
* not the first person from a household to enroll in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Well-Being (Psychological Flourishing) | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  Well-being will be self reported using an 8-item measure from Diener et al., 2010

SECONDARY OUTCOMES:
Life Satisfaction | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  1-item question by Fleeson, 2004
Stress | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  1 Item Statistics Canada Stress Question from the Canadian Community Health Survey (2012)
Depression | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  10 Item Center for Epidemiologic Studies Depression Scale (CES-D) via Andresen et al., 1994
Resilience | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  6 item Brief Resilience Scale by Smith et al., 2008
Social Identification | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  items adapted from the 4-item scale by Doosje et al., 1995
Social and Emotional Lonliness | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  11-item scale by De Jong Gierveld et al., 2006
Chronic Illness (Physical Health) | Baseline (Week 0)
  question by Charles et al., 2006 adapted from Larsen et al., 1991
Weekly Somatic Symptoms (Physical Health) | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  question by Charles et al., 2006 adapted from Marmot et al., 1997
Leisure-time physical activity | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  modified version of the Leisure Score Index (LSI; Courneya, Jones, Rhodes, & Blanchard, 2004) that has been applied to Godin's Leisure Time Exercise Questionnaire (GLTEQ; Godin & Shepard, 1985).
Alcohol Habits | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  3-item measure for alcohol consumption from CDC Behavioral Risk Factor Surveillance System Survey Questionnaire, 1984-2019
Physical Adherence | Looked at each day of the week for 12 weeks to see if a session was attended
  Objective measure of attendance in online sessions (interventions conditions only)
Affective Attitudes | Baseline (Week 0), Week 2, Week 4, Week 6, Week 8, Week 10, Follow-up (Week 12)
  3 semantic differential items toward physical activity using scale by Azjen, 2006
Demographics | Baseline only (Week 0)
  Items addressing sex/gender, age, ethnicity, sexual orientation, chronic conditions, smoking behaviour, height, weight, education level, household income level, employment status, marital status, and living situation (i.e., alone vs. others).

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The protocol for this study will be available on Open Science Framework (after 4 months to allow for study completion). The Statistical Analysis Plan will also be available on Open Science Framework. The Consent form is freely available if requested from the Primary Investigator (PI: Beauchamp, M.).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available from this trial 1 year after completion of the study. The data will remain available indefinitely.
Access Criteria: The nature of the request for sharing access will be reviewed by the PI (Beauchamp, M) and the data management team. Data will be shared via secure platforms (Redcap). Contact for data access can be done through personal communications (e.g., email) with PI Beauchamp.
URL: https://osf.io/xw9gm

REFERENCES:
- [Background] Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi, D. W., Oishi, S., & Biswas-Diener, R. (2010). New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social indicators research, 97(2), 143-156.
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] De Jong Gierveld, J, Tilburg, TV. A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Research on Aging. 2006; 28(5): 582-598.
- [Background] Charles, S.T. & Almeida, D.M. Daily reports of symptoms and negative affect: Not all symptoms are the same. Psychology & Health. 2006; 21(1): 1-17
- [Background] Fleeson, W. (2004). The quality of American life at the end of the century. In O. G. Brim, C. D. Ryff, & R. C. Kessler (Eds.), How healthy are we? A national study of wellbeing at midlife. Chicago: University of Chicago Press.
- [Background] Statistics Canada (2012), Canada Canadian Community Health Survey. Share File, Knowledge Management and Reporting Branch, Ontario MOHLTC
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Doosje, B., Ellemers, N., Spears, R. (1995) Perceived intragroup variability as a function of group status and identification. Journal of Experimental Social Psychology 31(5): 410-436.
- [Background] Larsen RJ, Kasimatis M. Day-to-day physical symptoms: individual differences in the occurrence, duration, and emotional concomitants of minor daily illnesses. J Pers. 1991 Sep;59(3):387-423. doi: 10.1111/j.1467-6494.1991.tb00254.x. PMID 1960638
- [Background] Marmot M, Ryff CD, Bumpass LL, Shipley M, Marks NF. Social inequalities in health: next questions and converging evidence. Soc Sci Med. 1997 Mar;44(6):901-10. doi: 10.1016/s0277-9536(96)00194-3. PMID 9080570
- [Background] Courneya KS, Jones LW, Rhodes RE, Blanchard CM. Effects of different combinations of intensity categories on self-reported exercise. Res Q Exerc Sport. 2004 Dec;75(4):429-33. doi: 10.1080/02701367.2004.10609176. No abstract available. PMID 15673042
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Centers for Disease Control and Prevention (CDC). (1984 - 2019). Behavioral Risk Factor Surveillance System Survey Questionnaire. Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention.
- [Background] Ajzen, I. (2006). Constructing a TPB questionnaire: Conceptual and methodological considerations. Retrieved from https://pdfs.semanticscholar.org/0574/b20bd58130dd5a961f1a2db10fd1fcbae95d.pdf
- [Derived] Beauchamp MR, Hulteen RM, Ruissen GR, Liu Y, Rhodes RE, Wierts CM, Waldhauser KJ, Harden SH, Puterman E. Online-Delivered Group and Personal Exercise Programs to Support Low Active Older Adults' Mental Health During the COVID-19 Pandemic: Randomized Controlled Trial. J Med Internet Res. 2021 Jul 30;23(7):e30709. doi: 10.2196/30709. PMID 34328433